CLINICAL TRIAL: NCT05286047
Title: Effects of Oral Bifidobacterium Longum CCFM1029 on Atopic Dermatitis in Infant
Brief Title: Probiotic on Atopic Dermatitis in Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glac Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hsieh-Hsun Ho, R&D Director, Glac Biotech Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH-2021001
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Probiotics; Intestinal flora; Allergic diseases
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium longum CCFM1029 (Experimental)
  Interventions: Dietary Supplement: Bifidobacterium longum CCFM1029
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum CCFM1029 — Subjects take one capsule containing Bifidobacterium longum CCFM1029 daily at bedtime.
  Arms: Bifidobacterium longum CCFM1029
Dietary Supplement: Placebo — Subjects take one capsule containing maltodextrin daily at bedtime.
  Arms: Placebo

SUMMARY:
The clinical trial will be carried out in China Medical University Hospital. The overall plan is a double-blind trial. All recruited 3 months-3 years old atopic dermatitis (AD) patients are divided into two groups, 50 in each group and 100 in two groups. The two groups are placebo and Bifidobacterium longum CCFM1029. The entire evaluation plan lasts for 3 months. The number of probiotic bacteria is 5 billion per capsule, and the number of bacteria taken by the subjects is 5 billion per day (one capsule before bed each day). During the planning period, the eczema area and severity index (EASI) score of the patient's dermatitis was evaluated every month, and the score differences of dermatitis before and after taking probiotics was observed. In addition, subjects must perform two fecal samplings before and after the trial, and the isolated DNA was analyzed using the next-generation high-throughput sequencing method (NGS) for subject fecal flora changes. Comparing the two groups before and after taking the capsule, whether the intestinal flora changed. Statistical analysis of the relationship between changes in intestinal flora and the degree of AD. Through the above test, the investigators evaluated whether Bifidobacterium longum CCFM1029 can regulate the pediatric intestinal flora and relieve the inflammatory response in the body, thereby regulating atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were between 3 months and 3 years old.
* For patients diagnosed with atopic dermatitis by a professional physician and the EASI score is greater than 5, the type and frequency of drugs used during the experiment should be recorded.
* The subject's parents agree to join the trial and sign the informed consent form.

Exclusion Criteria:

* The patient who has a history of allergic reactions, or the use of other highly sensitive or contraindicated drugs (allergy to antibiotics or antipyretics).
* The patient who has taken oral immunosuppressants and systemic steroids within the past 2 weeks.
* The patient who has consumed probiotic-related products (including drops, lozenges, capsules, powder or yogurt) within the past 1 month.
* The patient who has participated in other clinical studies within the past 1 month.
* The patient who has received immunotherapy within the past 1 year.
* The patient who suffering from major diseases (with a IC card for severe illness), congenital diseases.
* The patient who is not suitable to participate in the trial as assessed by the professional physician.

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Changes in eczema area and severity index (EASI) scores. | Before and 3-month intervention.
  Changes in eczema area and severity index (EASI) scores were assessed before and 3 months of intervention. The minimum value is "0" and maximum value is "72", higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes in eczema area and severity index (EASI) scores. | After 1 month and 2 months of intervention.
  Changes in eczema area and severity index (EASI) scores were assessed after 1 month and 2 months of intervention. The minimum value is "0" and maximum value is "72", higher scores mean a worse outcome.
Changes in gut microbiota ratios. | Before and 3 months of intervention.
  Changes in gut microbiota ratios were assessed by NGS before and 3 months of intervention.
Changes in infants' dermatitis quality of life (IDQOL) index. | Before and 1-, 2- and 3-month intervention.
  Changes in infants' dermatitis quality of life (IDQOL) index were assessed by questionnaire before and 1-, 2- and 3-month intervention. The minimum value is "0" and maximum value is "30", higher scores mean a worse outcome.
Changes in dermatitis family impact (DFI) scores. | Before and 1-, 2- and 3-month intervention.
  Changes in dermatitis family impact (DFI) scores were assessed by questionnaire before and 1-, 2- and 3-months intervention. The minimum value is "0" and maximum value is "30", higher scores mean a worse outcome.
Changes in subjects' frequency of medicine use from questionnaires. | Before and 1-, 2- and 3-month intervention.
  Changes in subjects' frequency of medicine use were assessed from questionnaire before and 1-, 2- and 3-months intervention. When subjects returned to the clinic, the average daily medicine use over the past month is asked by a professional physician.

CONTACTS AND LOCATIONS:
Locations (1):
- Glac Biotech Co., Ltd., Tainan, Taiwan